CLINICAL TRIAL: NCT07037888
Title: Efficacy of Ketorolac for Postoperative Pain Management in Hip Arthroscopy: A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Ketorolac for Postoperative Pain Management in Hip Arthroscopy: A Prospective Double-Blinded Randomized Controlled Trial
Acronym: Keto
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Thomas Lynch, Sports Medicine Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16671
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Femoracetabular Impingement; Hip Arthroscopy
Keywords: Sports Medicine; Hip Arthroscopy; FAI; Opioids; Ketorolac; Multi-modal pain
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Ketorolac; Omeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The standard of care/control pain protocol
  Interventions: Drug: Control (Standard treatment)
- Ketorolac (Active Comparator): Intra-operative IV and Oral doses of Ketorolac plus Standard of care
  Interventions: Drug: Ketorolac; Drug: Control (Standard treatment); Drug: Omeprazole

INTERVENTIONS:
Drug: Ketorolac — IV ketorolac intraoperative loading dose Ketorolac 10mg 1 tablet q6hrs to start on POD0
  Arms: Ketorolac
Drug: Control (Standard treatment) — hydrocodone-acetaminophen 5mg/325mg 1 tablet q6hrs PRN to start on POD0 30 tablets
Drug: Control (Standard treatment) — indomethacin 75mg 1 tablet QD to start on POD0 10 tablets
Drug: Control (Standard treatment) — diazepam 5mg 1-2 tablets q8hrs PRN to start on POD0 15 tablets
Drug: Omeprazole — 20 mg qd
  Arms: Ketorolac

SUMMARY:
The goal of this clinical trial is to learn whether the medication ketorolac can help manage pain after hip arthroscopy as well or better than the standard opioid-based pain medications. This study focuses on adult patients (over 18 years old) undergoing hip arthroscopy at Henry Ford Health System in Detroit, Michigan. Both men and women are included, and all participants must be able to consent and communicate in English.

The main questions it aims to answer are:

Can ketorolac help control pain as effectively or better than opioids after hip arthroscopy?

Will ketorolac use reduce the amount of opioid medication needed after surgery?

Researchers will compare the group receiving ketorolac to the group receiving standard opioid pain medications to see if ketorolac reduces pain and opioid use after surgery.

Participants will:

Be randomly assigned to one of two groups:

The control group, which receives the current standard pain management protocol (hydrocodone-acetaminophen and diazepam)

The experimental group, which receives the same protocol plus ketorolac and a stomach-protecting medication (omeprazole)

Receive their assigned pain medications after hip arthroscopy

Be asked to:

Take the prescribed medications after discharge

Complete a pain journal for 5 days following surgery, documenting pain levels and any side effects

Complete follow-up surveys and assessments at 2 weeks, 6 weeks, and 3 months after surgery

The main measurement researchers will use is the Visual Analog Scale (VAS) for pain on post-operative day 4. Additional measures include how many narcotic pills are used and results from PROMIS physical function and pain interference scores.

The hope is that ketorolac will provide equal or better pain control without the risks of addiction and side effects associated with opioid medications. If successful, this approach could offer a safer alternative for managing pain after hip arthroscopy. Participants may personally benefit by having effective pain relief with fewer risks, and future patients could benefit from improved pain management options.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip arthroscopy over the age of 18 with Dr. T. Sean Lynch
* Diagnosis of femoroacetabular impingement (FAI)

Exclusion Criteria:

* Patients with inability to consent and/or do not speak English
* Patients with conditions contraindicated with NSAIDs (medication allergy, peptic ulcer disease, bleeding diathesis, and renal disease)
* Patients with history of drug and alcohol use disorder
* Patients with chronic analgesia (filled two opioid prescriptions within 6 months of the surgery)
* Patients with psychotropic medication usage
* Patients who take pentoxifylline, probonecid, aspirin, and/or NSAIDs who cannot stop taking it for the study
* Patients who are not discharged same day after surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 5 days
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine.

SECONDARY OUTCOMES:
PROMOIS- PF | 2 weeks, 6 weeks, 3 months
  a patient-reported outcome measure that assesses an individual's self-reported capability to perform physical activities, including both basic activities of daily living (ADLs) and instrumental activities of daily living (IADLs)
PROMOIS- PI | 2 weeks, 6 weeks, 3 months
  a patient-reported outcome measure that assesses the extent to which pain hinders a person's engagement in various activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

REFERENCES:
- [Background] Bloom DA, Kirby DJ, Thompson K, Baron SL, Chee C, Youm T. Effect of Acetaminophen on Postoperative Percocet Use In Hip Arthroscopy: A Randomized Controlled Trial. Arthroscopy. 2021 Feb;37(2):530-536. doi: 10.1016/j.arthro.2020.09.046. Epub 2020 Oct 10. PMID 33045334
- [Background] Moutzouros V, Jildeh TR, Tramer JS, Meta F, Kuhlmann N, Cross A, Okoroha KR. Can We Eliminate Opioids After Anterior Cruciate Ligament Reconstruction? A Prospective, Randomized Controlled Trial. Am J Sports Med. 2021 Dec;49(14):3794-3801. doi: 10.1177/03635465211045394. Epub 2021 Oct 20. PMID 34668795
- [Background] Jildeh TR, Abbas MJ, Hasan L, Moutzouros V, Okoroha KR. Multimodal Nonopioid Pain Protocol Provides Better or Equivalent Pain Control Compared to Opioid Analgesia Following Arthroscopic Rotator Cuff Surgery: A Prospective Randomized Controlled Trial. Arthroscopy. 2022 Apr;38(4):1077-1085. doi: 10.1016/j.arthro.2021.11.028. Epub 2021 Nov 25. PMID 34838987
- [Background] LaPorte C, Rahl MD, Ayeni OR, Menge TJ. Postoperative Pain Management Strategies in Hip Arthroscopy. Curr Rev Musculoskelet Med. 2019 Dec;12(4):479-485. doi: 10.1007/s12178-019-09579-x. PMID 31650392
- [Background] Kahlenberg CA, Patel RM, Knesek M, Tjong VK, Sonn K, Terry MA. Efficacy of Celecoxib for Early Postoperative Pain Management in Hip Arthroscopy: A Prospective Randomized Placebo-Controlled Study. Arthroscopy. 2017 Jun;33(6):1180-1185. doi: 10.1016/j.arthro.2017.01.016. Epub 2017 Mar 1. PMID 28258773
- [Background] Beck EC, Nwachukwu BU, Jan K, Krivicich LM, Chahla J, Fu MC, Nho SJ. The Effect of Postoperative Opioid Prescription Refills on Achieving Meaningful Clinical Outcomes After Hip Arthroscopy for Femoroacetabular Impingement Syndrome. Arthroscopy. 2020 Jun;36(6):1599-1607. doi: 10.1016/j.arthro.2020.02.007. Epub 2020 Feb 14. PMID 32061972
- [Background] Jamil M, Dandachli W, Noordin S, Witt J. Hip arthroscopy: Indications, outcomes and complications. Int J Surg. 2018 Jun;54(Pt B):341-344. doi: 10.1016/j.ijsu.2017.08.557. Epub 2017 Aug 18. PMID 28823795